CLINICAL TRIAL: NCT02437344
Title: Glutamatergic Modulation to Facilitate Naltrexone Initiation in Opioid Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elias Dakwar, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #7057
Record Dates: First submitted 2015-04-26; First posted 2015-05-07 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — GluN2C-2D antagonist UBP145; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CI-581aa (Experimental): CI-581aa will be administered 24 hours after last opioid use, and followed by naltrexone dosing
  Interventions: Drug: CI-581aa; Drug: Naltrexone titration and XR-NTX initiation

INTERVENTIONS:
Drug: CI-581aa — 92 minute infusion of CI-581aa
  Other Names: NMDA antagonist
Drug: Naltrexone titration and XR-NTX initiation — participants will be provided a titration of naltrexone that culminates in the injection of XR-NTX
  Other Names: naltrexone

SUMMARY:
Opioid dependence is a substantial problem associated with significant morbidity and mortality. Extended-release naltrexone has been found effective at reducing opioid use and maintaining abstinence, but its use has been limited by the difficulties encountered with treatment initiation, which involves detoxification from opioids and oral naltrexone titration. Improving the likelihood of a successful transition to naltrexone is therefore an important public health goal.

N-methyl-D-aspartate receptor (NMDA) antagonism has been found to alleviate the signs and symptoms of withdrawal from opioids, as well as to address adaptations associated with chronic opioid use, such as opioid-induced hyperalgesia (increased pain sensitivity). These benefits may persist for at least 72 hours after a single dose. NMDA antagonism may therefore facilitate a rapid transition to naltrexone by reducing discomfort, improving motivation, and ameliorating adaptations associated with drug dependence, such as craving and arousal.

The purpose of this trial is to assess the feasibility of NMDA antagonist-assisted naltrexone initiation in opioid dependent individuals. After administration of extended-release naltrexone, participants will be followed for 4 weeks, and transitioned to appropriate care subsequently (oral naltrexone, extended-release naltrexone).

ELIGIBILITY:
Inclusion Criteria:

1. Active opioid dependence, with at least one positive utox result; no history of opioid overdose; and not currently using methadone or buprenorphine
2. Physically healthy
3. No adverse reactions to study medications
4. 21-60 years of age
5. Capacity to consent and comply with study procedures
6. Seeking treatment

Exclusion Criteria:

1. Meets DSM IV criteria for current major depression, bipolar disorder, schizophrenia, any psychotic illness, including substance-induced psychosis, and current substance-induced mood disorder with HAMD > 12.
2. Physiological dependence on another substance requiring medical management, such as alcohol or benzodiazepines, excluding caffeine, nicotine, and cannabis
3. Pregnant or interested in becoming pregnant
4. Delirium, Dementia, Amnesia, Cognitive Disorders, or dissociative disorders
5. Current suicide risk or a history of suicide attempt within the past 2 years
6. On psychotropic or other medication whose effect could be disrupted by participation in the study
7. Recent history of significant violence (past 2 years).
8. Heart disease as indicated by history, abnormal ECG, previous cardiac surgery.
9. Unstable physical disorders which might make participation hazardous such as end-stage AIDS, hypertension (>140/90), anemia, active hepatitis or other liver disease (transaminase levels < 2 X the upper limit of normal will be considered acceptable), or untreated diabetes
10. Previous history of CI-581 abuse, and/or a history of adverse reaction/experience wtih prior exposure to CI-581 or benzodiazepines
11. BMI > 35, or a history of unmanaged obstructive sleep apnea
12. First degree relative with a psychotic disorder (bipolar disorder with psychotic features, schizophrenia, schizoaffective disorder, or psychosis NOS)
13. History of opioid overdose over the past 2 years requiring medical intervention
14. Currently using methadone or buprenorphine

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elias Dakwar, MD, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CI-581aa
Started | 16
Completed | 15
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | CI-581aa
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16
baseline opioid use (morphine equivalents) [Mean (Standard Deviation); unit: morphine eq, in mg] | 297.7 (113.2)

OUTCOME MEASURES:

1. Primary Outcome: Successful Naltrexone Initiation
Description: The proportion of participants enrolled in the trial and receiving the infusion to receive XR-NTX
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CI-581aa
Number analyzed (Participants) | 12
Participants | 11

2. Secondary Outcome: Withdrawal: Subjective Opioid Withdrawal Scale (SOWS) Scores at Baseline and Administered Subsequently
Description: Subjective Opioid Withdrawal Scale (SOWS) is a scale out of 64 points assessing withdrawal severity that is administered serially, every several hours, over the course of the naltrexone initiation. The questionnaire assesses symptoms that the patient rates on a scale of 0 (not at all) to 4 (extremely). The difference in total (sum) scores between baseline and end-of-induction will be reported. Scores range from 0 to 64.
Time Frame: 4 days
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CI-581aa
Number analyzed (Participants) | 12
units on a scale | 34 (7)

ADVERSE EVENTS:
Time Frame: 2 months, from treatment entry through the 1 month follow-up.
Description: It does not differ.
Arm/Group | CI-581aa
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No